CLINICAL TRIAL: NCT00252109
Title: New Orleans AIDS Task Force Adopting and Demonstrating the Adaptation of Prevention Techniques (ADAPT) With Popular Opinion Leader (POL)
Brief Title: ADAPT-POL New Orleans: Adaptation of Prevention Techniques With Popular Opinion Leader
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CDC-NCHSTP-U65/CCU623818; U65/CCU623818-01-1 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: HIV Infections
Keywords: HIV; Seropositive; MSM; African American; Popular Opinion Leader
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Popular Opinion Leader — Popular opinion leaders of social networks are identified and attend 4 sessions to prepare them to have casual conversations with persons in the social networks that are meant to shift social norms to embrace safer behaviors (e.g., increased condom use, fewer sexual partners)
  Other Names: Adapted POL intervention also known locally as SouthPOL+.

SUMMARY:
Adopting and Demonstrating the Adaptation of Prevention Techniques (ADAPT) is a supplement to the Centers for Disease Control and Prevention (CDC) Community Based Organization Program Announcement 04064 (PA 04064). The purpose of ADAPT is to improve the understanding of the processes needed for adapting evidence-based behavioral interventions to fit new conditions or populations and to pilot the CDC-developed adaptation guidance. The ADAPT project responds to concerns from the field that existing interventions do not address the HIV prevention needs of their specific population. This project seeks to develop guidance for agencies to engage in the evidence-based adaptation of interventions previously shown to be effective in evaluation settings for use in real world applications.

The New Orleans AIDS Task Force (NO/AIDS) is one of five grantees funded to use the adaptation guidance to adapt an intervention packaged by the CDC's Replicating Effective Programs and disseminated by CDC's Diffusion of Effective Behavioral Interventions. The agency will adapt Jeff Kelly's Popular Opinion Leader (POL) intervention (Kelly, 2004; Kelly et al., 1991) for use in Internet venues with seropositive men who identify ethnically/racially as other than White/Caucasian who have sex with other men (men who have sex with men [MSM] of color).

Kelly's POL intervention is a community-level, evidence-based HIV prevention intervention that originally targeted gay and bisexual men in smaller cities throughout the United States. Kelly's intervention seeks to identify and enlist the support of well-known and well-liked opinion leaders to take on risk reduction advocacy roles. Opinion leaders attend sessions to learn how to engage in risk reduction conversations with people in their own social networks. The opinion leaders help to reshape social norms to encourage safer sex by helping to create a social environment in which MSM feel comfortable and empowered to make decisions to avoid high-risk sexual behaviors.

DETAILED DESCRIPTION:
In 2000, NO/AIDS was funded by the CDC to conduct community mobilization. Two components of that program were Kelly's POL and outreach in Internet chat rooms. Kelly's POL targeted traditional venues frequented by MSM, such as gay bars. Online outreach in chat rooms was modeled after standard street outreach, where outreach workers provide HIV/AIDS, sexually transmitted disease and risk reduction information and referrals. Since the agency started online outreach, the Internet has continued to grow and it has become a mainstream venue for MSM to seek sexual partners online while maintaining their anonymity (Benotsch et al., 2002; Bull et al., 2001). With this trend, the agency realized that the online MSM community needed to be targeted by multiple behavior change interventions comparable to those implemented in other at risk venues. The agency included implementation of Kelly's POL online in chat rooms frequented by MSM as one of the interventions to be funded through the CDC's PA 04064 (the parent grant). As of August 2004, the agency has been funded under the parent grant to conduct Kelly's POL online in chat rooms that serve New Orleans, Louisiana, and the Southeastern U.S. region. This parent grant project shall be referred to as South POL. Supplemental PA 04064 funding for ADAPT will be used to further adapt South POL to target seropositive MSM of color. The supplement grant project shall be referred to as South POL+.

The South POL+ intervention has three main goals: first, to adapt the intervention for use with adult seropositive MSM of color based on formative evaluation findings; second, to evaluate and monitor the process of adapting the intervention utilizing the CDC-developed Adaptation Guidance; and third, to conduct implementation monitoring and evaluation and evaluation of the implementation of the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive
* Men who have sex with other men
* African American
* At least 18 years of age
* Report having sexual contact with a man (any type of sexual contact in which either partner achieved orgasm) within the last year
* Those who frequent viable venues for recruiting pre-and post-implementation questionnaire respondents

Exclusion Criteria:

* MSM who are not willing to identify themselves to study staff as seropositive Hispanic MSM may be excluded.
* Those under 18 years of age will be excluded from participation due to the study design precluding direct applicability of hypotheses and intervention to both adults and children due to different cognitive development, HIV prevalence levels, and social networks.
* Serious mental illness which makes the individual unsuitable for participation
* Under the influence of drugs or alcohol which makes the individual unsuitable for participation
* Anyone who does not meet the inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men who have sex with men (MSM) of color who access Websites and chat rooms primarily frequented by MSM in the New Orleans, LA area.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2004-07; Primary Completion 2007-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Qualitative data collected during online focus groups to discuss risky sexual behavior engaged in by men who have sex with men (MSM) of color and access online venues primarily frequented by MSM in the New Orleans LA area. | Fall/winter 2006

SECONDARY OUTCOMES:
Development of Popular Opinion Leader behavioral HIV prevention intervention materials adapted for use online use with men who have sex with men (MSM) of color and who access online venues primarily frequented by MSM in the New Orleans LA area. | Spring 2007

CONTACTS AND LOCATIONS:
Overall Officials: Vel S. McKleroy, MPH, BSW, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- New Orleans AIDS Task Force, New Orleans, Louisiana, United States